CLINICAL TRIAL: NCT06333652
Title: Clinical Trial on the Use of Ravulizumab in Pregnancies Complicated by Severe Hypertensive Disorders
Brief Title: Ravulizumab in Pregnancies Complicated by Severe Hypertensive Disorders
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Maria Lourdes Gonzalez Suarez, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-009239
Record Dates: First submitted 2024-03-20; First posted 2024-03-27 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Preeclampsia
Keywords: Hemolysis; Elevated Liver enzymes; Low Platelets
MeSH Terms: conditions — Pre-Eclampsia; Hemolysis | interventions — ravulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Revulizumab Treatment (Experimental): Subjects will receive an single-dose infusion of Ravulizumab.
  Interventions: Drug: Ravulizumab

INTERVENTIONS:
Drug: Ravulizumab — Intravenous infusion 100 mg/ml
  Other Names: Ultomiris

SUMMARY:
The researchers are testing a medication named ravulizumab for the treatment of severe preeclampsia and Hemolysis, Elevated Liver enzymes, Low Platelets (HELLP) syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with < 34 0/7 weeks of gestation.
* Individuals with severe preeclampsia or HELLP features.

Exclusion Criteria:

* Pregnant female patients presenting with disseminated intravascular coagulopathy (DIC).
* Individuals with non-reassuring fetal status requiring delivery, non-viable fetuses, previable pregnancy (<23 0/7 weeks gestation), stroke, in utero fetal demise, known atypical hemolytic uremic syndrome, familial or acquired thrombocytopenia purpura, paroxysmal nocturnal hemoglobinuria, allergy to Ravulizumab, inability or unwillingness to sign informed consent.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Alternative Complement Pathway Biomarkers at time of delivery | Baseline
  Concentration in serum of biomarkers: sMAC, Bb, and C5 at time of delivery

SECONDARY OUTCOMES:
Pregnancy duration | Approximately 40 weeks
  Length of pregnancy measured in number of weeks.
Clinical biomarkers of severe features of preeclampsia and HELLP syndrome | 72 hours after Ravulizumab infusion
  Concentration of clinical biomarkers in serum: creatinine, AST, ALT, LDH and platelets
Hospitalization length in the postpartum period | Approximately 3-5 days, it may vary
  Length of hospital stay measured in number of days in hospital stay (peripartum period)
Meningococcal infection after use of ravulizumab | 72 hours up to 3 weeks after Ravulizumab infusion
  Number of participants to present a meningococcal infection after use of Ravulizumab

CONTACTS AND LOCATIONS:
Overall Officials: Maria Lourdes Gonzalez Suarez, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials